CLINICAL TRIAL: NCT00115414
Title: A Randomized, Double-Blind, Phase 2 Study Evaluating the Safety of Same Day Versus Next Day Administration of Pegfilgrastim With Docetaxel, Doxorubicin, and Cyclophosphamide (TAC) in Women With Breast Cancer
Brief Title: Same Day Dosing of Pegfilgrastim in Breast Cancer Patients Undergoing Chemotherapy (TAC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020778
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Breast Cancer; Fever; Neutropenia
Keywords: Neulasta®; Chemotherapy; TAC; Amgen
MeSH Terms: conditions — Breast Neoplasms; Fever; Neutropenia | interventions — pegfilgrastim; Docetaxel; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: pegfilgrastim
Drug: docetaxel
Drug: doxorubicin
Drug: cyclophosphamide

SUMMARY:
The purpose of this study is to provide data on the safety and efficacy of pegfilgrastim when administered on the same day versus the next day of chemotherapy, as measured by the duration of grade 4 neutropenia.

ELIGIBILITY:
Inclusion Criteria: - Breast cancer, previously untreated Exclusion Criteria: - Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, antiviral) within 72 hours of chemotherapy - Prior malignancy within the last 5 years, with the exception of surgically cured basal/squamous skin cell carcinoma, ductal carcinoma in situ of the breast and/or carcinoma of the cervix in situ - History of impaired cardiac status (e.g., severe heart disease, cardiomyopathy or congestive heart failure) - Major surgery within 2 weeks prior to randomization - Previous exposure to cytokines within two weeks prior - Concurrent use of other investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Neutropenia

SECONDARY OUTCOMES:
Neutropenia
Disease Response
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20020778.pdf